CLINICAL TRIAL: NCT02748967
Title: Randomized, Double-Blind, Placebo-controlled Phase 1 Study in Healthy Japanese Adult Subjects to Evaluate the Safety and Immunogenicity of Different Doses of JNJ-63871860
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Different Doses of ExPEC4V (JNJ-63871860) in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108139; 63871860BAC1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Healthy; ExPEC4V; JNJ-63871860; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Participants with age (greater than or equal to [>=] 20 to less than [<] 50 years) will receive single dose of 0.5 milliliter (mL) of ExPEC4V (4:4:4:4) or placebo on Day 1.
  Interventions: Drug: ExPEC4V; Drug: Placebo
- Group 2 (Experimental): Participants with age >= 20 to < 50 will receive single dose of 0.5 mL of ExPEC4V (8:8:8:8) or placebo on Day 1.
  Interventions: Drug: ExPEC4V; Drug: Placebo
- Group 3 (Experimental): Participants with age >= 20 to < 50 will receive single dose of 0.5 mL of ExPEC4V (16:16:16:16) or placebo on Day 1.
  Interventions: Drug: ExPEC4V; Drug: Placebo
- Group 4 (Experimental): Participants with age greater than or equal to [>=] 50 will receive single dose of 0.5 mL of ExPEC4V (4:4:4:4) or placebo on Day 1.
  Interventions: Drug: ExPEC4V; Drug: Placebo
- Group 5 (Experimental): Participants with age >= 50 will receive single dose of 0.5 mL of ExPEC4V (8:8:8:8) or placebo on Day 1.
  Interventions: Drug: ExPEC4V; Drug: Placebo
- Group 6 (Experimental): Participants with age >= 50 will receive single dose of 0.5 mL of ExPEC4V (16:16:16:16) or placebo on Day 1.
  Interventions: Drug: ExPEC4V; Drug: Placebo

INTERVENTIONS:
Drug: ExPEC4V — Participant will receive single dose 0.5 ml of ExPEC4V as intramuscular injection on Day 1.
  Other Names: JNJ-63871860
Drug: Placebo — Participant will receive single dose of Placebo on Day 1.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of different doses of ExPEC4V (JNJ-63871860) in healthy Japanese participants greater than or equal to [> =] 20 years of age.

DETAILED DESCRIPTION:
This is a Phase 1 double-blind (neither the Investigator nor the participant know the treatment), randomized (the study medication is assigned by chance), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study) parallel group, single center study in healthy Japanese participants aged greater than or equal to [> =] 20 years. A target of approximately 48 participants will be enrolled that are stratified according to their age in 2 groups: 24 participants > = 20 to less than [<] 50 years of age and 24 participants > = 50 years of age. Both groups will be randomized to a single vaccination with 1 of the 3 study dose levels of ExPEC4V or placebo (vaccine buffer). Participants will be enrolled in a dose ascending approach. Blood samples will be drawn on Days 1 (prevaccination), 15 and 30 for the assessment of immunogenicity. The study duration per participant will be approximately 38 days (Screening period and postvaccination follow-up included). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of, and procedures required for the study and is willing to participate in the study
* Participant must be a man or woman greater than or equal to [> =] 20 years of age on the day of signing the ICF
* A female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction until at least 3 months after study vaccine administration. A male participant must agree not to donate sperm until at least 3 months after study vaccine administration
* Participant must have a body mass index (BMI: weight in kg divided by the square of height in meters) of less than or equal to [< =] 30.0 kg/m^2
* A male participant who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a double barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner uses occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

* Participant has a history of neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) within the past 5 years or a history of any hematological malignancy
* Participant has current or a history of autoimmune disease
* Participant has received an investigational drug (including investigational vaccines) within 90 days before vaccination in the study or is currently enrolled in an investigational study
* Participant has received treatment with immunoglobulins or blood products in the 4 months before vaccination in the study or any plans to receive such treatment during the study
* Participant has known or suspected congenital or acquired immunodeficiency (including leukemia, human immunodeficiency virus [HIV] seropositivity), has received immunosuppressive therapy (such as cyclosporine, anti-cancer chemotherapy, radiation therapy, or cytotoxic drugs) within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent) for more than 2 consecutive weeks within the past 3 months, or has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen (HBsAg) and hepatitis C antibody, respectively

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to follow-up (30 days)

SECONDARY OUTCOMES:
Antibody Levels Against the ExPEC4V Measured by an Enzyme-Linked Immunosorbent Assay (ELISA) | Up to Day 30
Antibody Levels Against the ExPEC4V Measured by Opsonophagocytic Killing (OPK) Assay | Up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukuoka, Japan